CLINICAL TRIAL: NCT04980859
Title: A Phase III, Single-arm Clinical Trial of Zebutinib Combined With Immunochemotherapy With Limited Course of Treatment for Newly Treated Chronic Lymphocytic Leukemia Patients Without 17p-
Brief Title: Zebutinib Combined With Immunochemotherapy in the Treat of Newly Treated CLL Patients Without 17p-/TP53 Mutation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Ru Feng, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL-NFH-202103
Record Dates: First submitted 2021-07-09; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zebutinib Combined With CIT arm (Experimental): Zebutinib Combined With FCR( under 60 years of age) or BR (over 60 years of age )
  Interventions: Drug: Zebutinib&BR or Zebutinib&FCR

INTERVENTIONS:
Drug: Zebutinib&BR or Zebutinib&FCR — Introduction period: Zebutinib 160 mg bid oral treatment for 3 months;Joint stage :6 sessions of Zebutinib FCR( under 60 years of age,Fludarabine 25 mg/m² Q3W, Cyclophosphamide 250 mg/m² Q3W,Rituximab 375 mg/m² Q3W) or BR (over 60 years of age, )(28 days and 1 cycle);Maintenance treatment: after the end of the combined phase, continue the treatment of zebutinib.

SUMMARY:
To investigate limited course of treatment of Zebutinib combined with immunochemotherapy for patients with newly treated chronic lymphocytic leukemia without 17p-/TP53 mutation

ELIGIBILITY:
Inclusion Criteria:

* CLL patients with indications for treatment according to iwCLL;
* CT/MRI shows measurable lesions;
* ECOG score is 0-2;
* No pregnancy plans during treatment

Exclusion Criteria:

* Richter transformation;
* 17p-/TP53 amplification ≥20% (FISH);
* Received steroids within 7 days before starting treatment;
* Have previously received treatments for chronic lymphocytic leukemia;
* Vaccine live attenuated vaccine within 4 weeks of randomization;
* Any life-threatening disease;
* Central nervous system leukemia;
* Apoplexy, history of intracranial hemorrhage;
* HIV or HCV or HBVpositive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
MRD conversion rate (minimal residual disease conversion rate) | 30 days
  minimal residual disease conversion rate

SECONDARY OUTCOMES:
OS (overall survival) | 3 years
  overall survival
PFS (progression-free survival) | 3 years
  progression-free survival

IPD SHARING:
Plan to Share IPD: No